CLINICAL TRIAL: NCT02287558
Title: A Phase I Single Arm Study to Assess the Safety and Efficacy of Pomalidomide in Patients With Bleeding Due to Hereditary Hemorrhagic Telangiectasia and Refractory Angiodysplasia
Brief Title: Pomalidomide in Hereditary Hemorrhagic Telangiectasia and Transfusion-Dependent Vascular Ectasia: a Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Keith McCrae, Director of Benign Hematology, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4Z14
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Idiopathic Vascular Ectasia
Keywords: HHT; CASE4Z14; Pomalidomide
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomalidomide (Experimental): Pomalidomide will be supplied as 1.0 mg, 2.0 mg, 3.0 mg and 4.0 mg capsules for oral administration. The principal investigator will determine whether intrapatient dose escalation is indicated based on the response of the patient's bleeding during the first 30 days of therapy. If dose escalation is indicated, pomalidomide will be increased by 1 mg/month at the investigator's discretion to a maximal dose of 5 mg/day.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide
  Other Names: Pomalyst; CC-4047; Imnovid

SUMMARY:
This study will evaluate patients > 18 years of age with transfusion-dependent gastrointestinal bleeding due to documented gastrointestinal vascular ectasia with or without concurrent hereditary hemorrhagic telangiectasia (HHT). This study will focus on documented bleeding sites in the small bowel, including the duodenum, jejunum and ileum. Eligible patients will have endoscopically-documented sites of vascular ectasia and will have required at least 4 units of blood transfusion or episodes of intravenous iron administration over the preceding four months.

DETAILED DESCRIPTION:
This is a single-arm, open-label study that will investigate the efficacy and safety profile of pomalidomide in patients with genetically-documented Hereditary Hemorrhagic Telangiectasia (defined by characteristic mutations in Eng, Alk-1 or Smad-4) or idiopathic vascular ectasia with no documented mutations, leading to refractory bleeding of the small bowel. This study will be limited to patients with documented bleeding from the small bowel, including the duodenum, jejunum or ileum. Eligible patients will be dependent on transfusion or intravenous iron therapy (requiring at least 4 units of blood transfusion or 4 iron infusions over the preceding 4 months) and will have endoscopically-confirmed areas of vascular ecstasia. Therapy for all eligible patients will be initiated with a 1 mg daily dose of pomalidomide. The principal investigator will determine whether intrapatient dose escalation is indicated based on the response of the patient's bleeding during the first 30 days of therapy. If dose escalation is indicated, pomalidomide will be increased at the investigator's discretion to a maximal dose of 5 mg/day. Cessation of GI bleeding will be defined as maintenance of stable hemoglobin without blood transfusion or intravenous iron therapy over a 4 week period. Once GI bleeding has ceased, patients will be maintained at a stable pomalidomide dose for an additional 4 months, and the dose then tapered by 1 mg per month, or until bleeding recurs. Patients will be followed for a total of six months post-therapy to determine whether the response is maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Transfusion of at least 4 units of blood and/or four doses of intravenous iron over the preceding four months.
3. Recurrent bleeding after at least one previous interventional endoscopic procedure
4. Platelet count ≥ 125,000/µl
5. WBC ≥ 4,000/µl
6. Normal prothrombin (PT) and activated partial thromboplastin time (aPTT)
7. Endoscopically-documented angiodysplasia and/or arteriovenous malformations involving the small bowel
8. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy.
9. Ability to understand and sign informed consent
10. All study participants must be registered into the mandatory POMALYST REMS™ program, and be willing and able to comply with the requirements of the POMALYST REMS™ program

Exclusion Criteria:

1. Pregnancy (must be excluded by two urine or serum tests for β-HCG in all women of child-bearing potential).

   Pregnancy Testing -Must follow pregnancy testing requirements as outlined in the POMALYST REMS™ program.
2. Breast feeding
3. Renal insufficiency, serum creatinine > 2.0 mg/dl
4. Hepatic insufficiency, bilirubin > 2.0 or transaminases > 3.0 x normal
5. Previous treatment with Thalidomide or other imid drugs within previous 12 months
6. History of prior thromboembolism with known thrombophilia
7. Peripheral neuropathy, as determined from neurologic consultation
8. Underlying hypoproliferative anemia (i.e. myelodysplasia)
9. Inherited or significant acquired coagulopathy (i.e. hemophilia, advanced liver disease)
10. Chronic aspirin, NSAID therapy, anticoagulation therapy or antiplatelet agents
11. Currently enrolled in other interventional trials
12. Known hypersensitivity to thalidomide or lenalidomide.
13. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, or similar drugs.
14. Anything that in the investigator's opinion is likely to interfere with completion of the study † A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Transfusion requirement measure | 8 months
  To compare the requirement for transfusion and intravenous iron administration in individual patients in the 4 month period before initiation of pomalidomide with that over a 4 month period following pomalidomide therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Keith McCrae, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States